CLINICAL TRIAL: NCT06737068
Title: Low Pressure Pneumoperitoneum Using AirSeal® for Reduction in Postoperative Shoulder Pain Following Robot Assisted Hiatal Hernia Repair: a Prospective Randomized Controlled Trial.
Brief Title: Low Pressure Pneumoperitoneum Using AirSeal® for Reduction in Postoperative Shoulder Pain Following Robot Assisted Hiatal Hernia Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2068123-1
Record Dates: First submitted 2024-11-19; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hernia, Hiatal; Pneumoperitoneum; Postoperative Pain; Shoulder Pain
MeSH Terms: conditions — Hernia, Hiatal; Pneumoperitoneum; Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low Pressure Pneumoperitoneum (8-10 mmHg) (Experimental): Elective robot assisted hiatal hernia repair with pneumoperitoneum pressures of 8-10 mmHg throughout the case
  Interventions: Procedure: Low pressure pneumoperitoneum (8-10mmHg) with AirSeal device
- Standard Pressure Pneumoperitoneum (13-15 mmHg) (Other): Elective robot assisted hiatal hernia repair with pneumoperitoneum pressures of 13-15 mmHg throughout the case
  Interventions: Procedure: Standard pressure pneumoperitoneum (13- 15 mmHg) with AirSeal device

INTERVENTIONS:
Procedure: Low pressure pneumoperitoneum (8-10mmHg) with AirSeal device — Elective robot assisted hiatal hernia repair with low pressure pneumoperitoneum (8-10mmHg) with AirSeal device
  Other Names: low pressure
  Arms: Low Pressure Pneumoperitoneum (8-10 mmHg)
Procedure: Standard pressure pneumoperitoneum (13- 15 mmHg) with AirSeal device — Elective robot assisted hiatal hernia repair with standard pressure pneumoperitoneum (13- 15 mmHg) with AirSeal device
  Other Names: standard pressure
  Arms: Standard Pressure Pneumoperitoneum (13-15 mmHg)

SUMMARY:
The goal of this clinical trial is to evaluate the incidence and severity of post-operative shoulder pain following elective robot-assisted hiatal hernia repair in hopes of reducing pain and associated costs as well as clinic and emergency department visits due to this pain. You will undergo standard robot-assisted hiatal hernia repair with the standard postoperative care. The only difference is that you may be selected for the group where lower pressures used to fill your abdomen with carbon dioxide will be used, and you will be asked to fill out logs regarding your pain postoperatively. You will have postoperative appointments that are standard following this procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective robot assisted hiatal hernia repair

Exclusion Criteria:

* patients less than 18 years of age
* conversion to open surgery
* BMI > 40
* history of abdominoplasty
* history of chronic pain and/or opioid dependence
* history of COPD and/or supplemental oxygen use
* pregnant patients
* incarcerated patients
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in post-operative shoulder pain | 1 week (on average)
  Percentage reduction in post-operative shoulder pain from POD#0 to ~1 week post-operative telephone appointment

SECONDARY OUTCOMES:
Severity of postoperative shoulder pain on POD #0 | 6 hours (on average)
  Severity of postoperative shoulder pain on POD #0 (recorded at nursing shift change ~7PM)
Severity of postoperative shoulder pain on POD #1 | 18 hours (on average)
  Severity of postoperative shoulder pain on POD #1 (when surgical team rounds ~6-8AM)
Severity of postoperative shoulder pain at ~1 week | 1 week (on average)
  Severity of postoperative shoulder pain at ~1 week post-operative telephone appointment
Severity of postoperative shoulder pain at ~2 weeks post-op | 2 weeks (on average)
  Severity of postoperative shoulder pain at ~2 week postoperative clinic visit measured by numeric pain rating scale and morphine milligram equivalents
length of hospital stay | through study completion, an average of 2 years
  length of hospital stay
readmission rates for shoulder pain | through study completion, an average of 2 years
  readmission rates for chief complaint of shoulder pain
number of postoperative clinic visits related to shoulder pain management | through study completion, an average of 2 years
  number of postoperative clinic visits related to shoulder pain management
discharge disposition | through study completion, an average of 2 years
  discharge disposition (home, SNF, rehab, etc)
standard vs extended narcotic regimen | through study completion, an average of 2 years
  standard vs extended (requiring refill) narcotic regimen
quality of life | 1 week (on average)
  quality of life assessed via EQ-5D-5L and EQ-VAS questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside University Health System, Moreno Valley, California, United States

REFERENCES:
- [Background] Luketina R, Luketina TLH, Antoniou SA, Kohler G, Konneker S, Manzenreiter L, Wundsam H, Koch OO, Knauer M, Emmanuel K. Prospective randomized controlled trial on comparison of standard CO2 pressure pneumoperitoneum insufflator versus AirSeal(R). Surg Endosc. 2021 Jul;35(7):3670-3678. doi: 10.1007/s00464-020-07846-4. Epub 2020 Aug 7. PMID 32767145
- [Background] Buda A, Di Martino G, Borghese M, Restaino S, Surace A, Puppo A, Paracchini S, Ferrari D, Perotto S, Novelli A, De Ponti E, Borghi C, Fanfani F, Fruscio R. Low-Pressure Laparoscopy Using the AirSeal System versus Standard Insufflation in Early-Stage Endometrial Cancer: A Multicenter, Retrospective Study (ARIEL Study). Healthcare (Basel). 2022 Mar 14;10(3):531. doi: 10.3390/healthcare10030531. PMID 35327010
- [Background] Yasir M, Mehta KS, Banday VH, Aiman A, Masood I, Iqbal B. Evaluation of post operative shoulder tip pain in low pressure versus standard pressure pneumoperitoneum during laparoscopic cholecystectomy. Surgeon. 2012 Apr;10(2):71-4. doi: 10.1016/j.surge.2011.02.003. Epub 2011 Mar 21. PMID 22385527
- [Background] Wallace DH, Serpell MG, Baxter JN, O'Dwyer PJ. Randomized trial of different insufflation pressures for laparoscopic cholecystectomy. Br J Surg. 1997 Apr;84(4):455-8. PMID 9112891
- [Background] Topcu HO, Cavkaytar S, Kokanali K, Guzel AI, Islimye M, Doganay M. A prospective randomized trial of postoperative pain following different insufflation pressures during gynecologic laparoscopy. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:81-5. doi: 10.1016/j.ejogrb.2014.09.003. Epub 2014 Sep 16. PMID 25265495
- [Background] Sroussi J, Elies A, Rigouzzo A, Louvet N, Mezzadri M, Fazel A, Benifla JL. Low pressure gynecological laparoscopy (7mmHg) with AirSeal(R) System versus a standard insufflation (15mmHg): A pilot study in 60 patients. J Gynecol Obstet Hum Reprod. 2017 Feb;46(2):155-158. doi: 10.1016/j.jogoh.2016.09.003. Epub 2017 Jan 30. PMID 28403972
- [Background] Saway JP, McCaul M, Mulekar MS, McMahon DP, Richards WO. Review of Outcomes of Low Verses Standard Pressure Pneumoperitoneum in Laparoscopic Surgery. Am Surg. 2022 Aug;88(8):1832-1837. doi: 10.1177/00031348221084956. Epub 2022 Apr 20. PMID 35442815
- [Background] Sarli L, Costi R, Sansebastiano G, Trivelli M, Roncoroni L. Prospective randomized trial of low-pressure pneumoperitoneum for reduction of shoulder-tip pain following laparoscopy. Br J Surg. 2000 Sep;87(9):1161-5. doi: 10.1046/j.1365-2168.2000.01507.x. PMID 10971421
- [Background] Joshipura VP, Haribhakti SP, Patel NR, Naik RP, Soni HN, Patel B, Bhavsar MS, Narwaria MB, Thakker R. A prospective randomized, controlled study comparing low pressure versus high pressure pneumoperitoneum during laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2009 Jun;19(3):234-40. doi: 10.1097/SLE.0b013e3181a97012. PMID 19542853
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] Gurusamy KS, Vaughan J, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 18;2014(3):CD006930. doi: 10.1002/14651858.CD006930.pub3. PMID 24639018
- [Background] Foley CE, Ryan E, Huang JQ. Less is more: clinical impact of decreasing pneumoperitoneum pressures during robotic surgery. J Robot Surg. 2021 Apr;15(2):299-307. doi: 10.1007/s11701-020-01104-4. Epub 2020 Jun 22. PMID 32572753
- [Background] O'Connor SC, Mallard M, Desai SS, Couto F, Gottlieb M, Ewing A, Cobb WS, Carbonell AM, Warren JA. Robotic Versus Laparoscopic Approach to Hiatal Hernia Repair: Results After 7 Years of Robotic Experience. Am Surg. 2020 Sep;86(9):1083-1087. doi: 10.1177/0003134820943547. Epub 2020 Aug 18. PMID 32809844
- See also: Related Info — https://www.conmed.com/en-us/products/airseal-and-insufflation